CLINICAL TRIAL: NCT06580392
Title: Cardiac Contractility Modulation (CCM) and Implementation of Guideline-Directed Medical Therapy in Patients With Heart Failure
Brief Title: CCM and Implementation of Guideline-Directed Medical Therapy in Patients With Heart Failure (Fix-GDMT-HF)
Status: Recruiting | Type: Observational
Sponsor: Impulse Dynamics (Industry)
Responsible Party: Sponsor
Other Study IDs: ID_CA_PRO_2105
Record Dates: First submitted 2024-08-28; First posted 2024-08-30 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Heart Failure
Keywords: Change in Quad medication score
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The primary objective of this study is to evaluate the impact of Cardiac Contractility Modulation (CCM) therapy on the initiation and up-titration of Guideline-Directed Medical Therapy (GDMT) in patients with heart failure (HF). This will be assessed by the change in Quad Medication Score (QMS) from baseline (pre-CCM) to 6-month following post-CCM device implant.

DETAILED DESCRIPTION:
Design Prospective, non-randomized, comparison analysis of medication use and dosing at pre/post CCM therapy. The Fix-GDMT-HF study aims to enroll up to 200 subjects (100 in Investigational Arm and up to 100 in Registry Arm). Subjects identified not eligible to participate in the investigational arm can participate in the registry arm.

Method

* Subjects with QMS ≤ 5, eGFR ≥15, diagnosed symptomatic heart failure and LVEF ≤40% will be enrolled after review and approval by a member of the steering committee. Eligible subjects will receive CCM therapy and be enrolled in the investigational arm of the study. Medication optimization(Med op#2) will be assessed after implantation(approx. 3month post implant), followed by evaluation of QMS and other endpoints at 6 and 12 months. A target of 100 patients will be enrolled in the investigational arm.
* After medical optimization (Med op# 1), if the patient has QMS > 5 or identified during SC review as not eligible to participate in investigational arm can participate in the registry arm. They will continue treatment guided by local practice (including potential CCM implant) with QMS assessment (and other data collection as patients in investigational arm) at 6- and 12-month visit. The registry arm will be restricted to 100 patients.

Endpoints

Primary Endpoint:

• Change in the Quad Medication Score (QMS) from baseline (pre-CCM) to 6-month follow-up (post-CCM) of the Optimizer device implant.

Secondary Endpoints:

* Change in loop diuretic dose from baseline to 6-month follow-up.
* Change in eGFR from baseline to 6-month follow-up.
* Change in SBP from baseline to 6-month follow-up.
* Adverse events (AEs) associated with CCM therapy.
* Change in HR among patients with concomitant cardiac rhythm management (CRM) devices.
* Percentage of patients achieving maximal/optimal GDMT following CCM therapy.
* GDMT adherence as measured by change in QMS score from 6 months (post-CCM) to 12 months (post-CCM).

Patients

Investigational arm - 100 subjects complete the study with 12- month of follow-up.

Registry arm - restricted to 100 subjects

Sites 10 sites in Germany & Italy. 10 sites in the USA.

Duration

The entire study is expected to take approximately 24 months or (until the target number of subjects has been reached), including the enrolment and follow-up periods.

ELIGIBILITY:
Inclusion Criteria:

1. Adults (≥18 years) diagnosed with symptomatic heart failure
2. Patients with Heart failure with reduced Ejection Fraction (HFrEF) where the Ejection Fraction (EF) is ≤40%

   - Historical LVEF assessed up to 6 months prior to consent by any modality can be used if available
3. Patients can have an active concomitant CRT device already - implanted provided the following criteria:

   * CRT device has been implanted >1 year
   * Patients are functional class NYHA III-IV

Exclusion Criteria:

1. Patients that are unlikely to adhere to medical therapy for reasons other than intolerance or contraindications.
2. Patients with a QMS score >5
3. eGFR <15
4. Patients with a concomitant CRT device that has already been implanted and deemed to be a responder
5. Patients with class I indication for a concomitant CRT device
6. Patients with significant comorbidities or conditions that may interfere with the study assessments
7. Patients with contraindications to CCM therapy or unable to undergo implantation
8. Severe stenotic valve disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subject selection will be based on specific inclusion and exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Change in Quad Medication Score | 6 month
  Change in the Quad Medication Score (QMS) from baseline (pre-CCM) to 6-month follow-up (post-CCM) of the Optimizer device implant

SECONDARY OUTCOMES:
Change in loop diuretic dose | 6-month
  Change in loop diuretic dose from baseline to 6-month follow-up.
Change in eGFR | 6-month
  Change in eGFR from baseline to 6-month follow-up
Change in SBP | 6-month
  Change in SBP from baseline to 6-month follow-up.
Adverse events (AEs) associated with CCM therapy. | 12-month
  Adverse events (AEs) associated with CCM therapy.
Percentage of patients achieving maximal/optimal GDMT following CCM therapy | 12-month
  Percentage of patients achieving maximal/optimal GDMT following CCM therapy
GDMT adherence as measured by change in QMS score | 12-month
  GDMT adherence as measured by change in QMS score from 6 months (post-CCM) to 12 months (post-CCM).

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Gemelli University Hospital, Rome, Italy
  - AO dei Colli - O.Monaldi, Napoli

IPD SHARING:
Plan to Share IPD: No